CLINICAL TRIAL: NCT01280370
Title: Prospective Evaluation of Laparoscopic and Open Hernia Repair: a Multicenter Cohort Study
Brief Title: Prospective Evaluation of Laparoscopic and Open Incisional Hernia Repair: a Multicenter Cohort Study
Acronym: IHR_SALTC
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 231/09
Record Dates: First submitted 2011-01-19; First posted 2011-01-20 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Incisional Hernia Repair
Keywords: Incisional hernia repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: 1.patients treated in a laparoscopic manner
- 2.: 2. patients treated in open operative manner
  Interventions: Procedure: Abdominal surgery

INTERVENTIONS:
Procedure: Abdominal surgery — intraoperative mesh implantation
  Groups: 2.

SUMMARY:
Nowadays incisional hernia are primarily repaired using prosthetic meshes. In Switzerland such meshes are mainly implanted via open or laparoscopic approach. The differential impact of these two types of surgical technique on recurrence rate will be investigated with this study.

With this multicenter cohort study the outcomes of laparoscopic and open incisional hernia repair will be investigated prospectively. Hernia recurrence is the main outcome measure.

Hypothesis:

Laparoscopic incisional hernia repair is associated with a lower recurrence rate compared to open incisional hernia repair.

DETAILED DESCRIPTION:
Background

Incisional hernia is a common long-term complication following abdominal surgery and is estimated to occur in 11-23% 1-3. Incisional hernia can be repaired by an open or by a laparoscopic approach. For incisional hernia prosthetic meshes are nowadays implanted for virtually all open and laparoscopic procedures.

The use of laparoscopy for the treatment of incisional hernia was first reported in 1993 by LeBlanc and Booth 4. Short term follow-up studies show that laparoscopic surgery is associated with decreased postoperative pain, reduced risks of surgical site infections due to minimal tissue dissection, a shorter length of hospital stay and a shorter overall recovery period 5-9.

Important long- term outcome parameters are recurrence rate and chronic pain 10,11. Recurrence after incisional hernia repair varies widely and ranges from 1% to 35% 1,3. Morbid obesity, a previous failed open repair, large defect size and postoperative complications are associated with an increased risk for recurrence 12. Heterogeneity of hernia size and follow-up further complicate comparison of the recurrence rate between different techniques. On average, 74% of recurrences occur within the first 3 years after initial repair 13. Series with an acceptable follow-up of at least 24 months report a recurrence rate in open and laparoscopic repair of approximately 10% 1. Currently, no well designed prospective study is available comparing the incidence of recurrence between open and laparoscopic incisional hernia repair.

Such variability of patients characteristics, surgical techniques and surgical skills are likely to confound a prospective randomized trial. Consequently, a cohort study is performed allowing each surgeon to perform the technique he is most familiar with.

The aim of this multicenter cohort study is to assess the incidence of recurrence 36 months after open and laparoscopic incisional hernia repair, performed in swiss hospitals.

Objective

All patients undergoing elective incisional hernia repair who meet the inclusion criteria (see below) are eligible for inclusion into the study. These patients will be informed about the details of the study preoperatively. After a patient has agreed to enroll into the study and has signed written informed consent, he/she will be advised to attend follow-up assessments according to the study plan.

Methods

All patients undergoing elective incisional hernia repair who meet the inclusion criteria (see below) are eligible for inclusion into the study. These patients will be informed about the details of the study preoperatively. After a patient has agreed to enroll into the study and has signed written informed consent, he/she will be advised to attend follow-up assessments according to the study plan.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Written informed consent
* Primary or recurrent incisional hernia

Exclusion Criteria

* Systemic or severe local infections
* Emergency procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing incisional hernia repair
Sampling Method: Non-Probability Sample
Enrollment: 371 (Actual)
Dates: Start 2010-09; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
recurrence rate | 36 months

SECONDARY OUTCOMES:
surgical site infections | 36 months
chronic pain | 36 months
length of hospital stay | 3 months
morbidity | 3 months
cosmetic results | 36 months
rigidity of the abdominal wall | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Guido Beldi, Prof. Dr. med., Principal Investigator — Berne, University Hospital, University of Berne, Switzerland
Locations (1):
- Dep. of Visceral and transplant surgery, Berne University Hospital, Bern, Switzerland